CLINICAL TRIAL: NCT06681246
Title: The Role of Microbiome in Recurrent Obesity Before and After Antibiotic/Placebo Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weizmann Institute of Science (Other)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0744-21-HMO
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic treatment (Experimental): intervention arm
  Interventions: Other: Antibiotic treatment
- Placebo (Placebo Comparator): placebo capsules administration
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Antibiotic treatment — 10 days of either antibiotics- Augmentin (amoxicillin+clauvonate), 875mg, 2 /day
  Arms: Antibiotic treatment
Other: Placebo — consist of a combination of agarose in normal saline/glycerol
  Arms: Placebo

SUMMARY:
This past century witnessed a significant increase in the prevalence of obesity. Successful weight loss maintenance is defined as losing at least 10% of the initial body weight and maintaining it for at least one year. However, keeping a low body weight is rarely maintained, as 80% of people who lost 10% of their body weight will return to their initial weight within a year. Although there is no agreement as to what contributes to the recurrent weight regain phenomenon (also known as 'weight cycling' or 'yo-yo diet'), it is strongly associated with the risk of developing metabolic risk factors and their complications, including heart disease and all-cause mortality. Altering the gut microbiota is one method to treat disease states associated with gut bacteria. Antibiotics consumption is known to influence host glycemic response through changes induced in microbiome composition and function. Therefore, it may be a possible pathway to jumpstart changes in the gut microbiota.

This study will determine whether microbiome modulation might be a possible future target against recurrent obesity in humans and whether orally administered antibiotic treatment post-weight loss might be an effective intervention to prevent weight regain.

DETAILED DESCRIPTION:
This is a placebo-controlled, double blinded interventional study evaluating the effect of antibiotic treatment in the prevention of weight regain after a successful weight loss intervention.

Volunteers will be recruited in the following ways: e-mail, and social media. Volunteers wishing to participate will be asked to complete a questionnaire regarding the aforementioned inclusion and exclusion criteria. Volunteers who qualify for the study will be invited to an introductory meeting at the Weizmann Institute of Science. The details of the experiment and potential risks or discomforts involved in it will be presented, after which the volunteers will sign an informed consent form. Volunteers will start the study and become active participants for a maximal duration of one year.

Samples collected for the study will be used for microbiota profiling (stool and oral), metabolomics (stool, blood) and for bomb calorimeter (stool).

The study will comprise of four parts:

1. Baseline - one week of profiling and screening.
2. Nutritional intervention - weight loss intervention which will be based on personalized hypocaloric diet restriction. Meetings will occur twice a month starting from the second week of the study for a three-month period.
3. Antibiotic treatment - 10 days of either antibiotics- Augmentin (amoxicillin+clauvonate), 875mg, 2 /day, or 10 days of placebo pills, 2/day.
4. Follow-up meetings - total follow up of 9 months after antibiotic/placebo treatment. Meetings will occur once a month for the first 3 months of the follow up period, and once every 3 months, afterwards.

ELIGIBILITY:
Inclusion Criteria:

* 28<BMI<35
* Age - 18-65
* Capable of working with a smartphone application

Exclusion Criteria:

* Consumption of antibiotics/probiotics/oral antifungals 2 months prior to the first day of the experiment.
* Pregnancy, fertility treatments, breastfeeding women six months prior to enrollment and during the study.
* Chronic disease, to the discretion of the study team (e.g. AIDS, Cushing syndrome, CKD, acromegaly etc.)
* Cancer and recent anticancer treatment
* Psychiatric disorders, to the discretion of the study team.
* Coagulation disorders
* IBD (inflammatory bowel diseases)
* Bariatric surgery.
* Eating disorders (Anorexia nervosa. Bulimia nervosa. Binge eating disorder, Night eating syndrome).
* Alcohol or substance abuse
* Weight loss attempts 6 months prior to the first day of the experiment - using weight loss medication.
* Drastic changes in nutritional habits six months prior to the first day of the study - to the discretion of the study team.
* Allergy to penicillin.
* Life threatening reaction after consumption of cephalosporins.
* History of CDI
* Liver disease
* History of serious unresolved diarrhea in response to antibiotic treatment to the discretion of the study doctor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
microbiome composition | 1 year
  using stool and oral samples
weight | 1 year
  weight (kg)

SECONDARY OUTCOMES:
glycemic response | 1 year
  continues glucose monitor (CGM)

CONTACTS AND LOCATIONS:
Overall Officials: Hila Elinav, Doctor, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Weizmann Institute of Science, Rehovot, Israel